CLINICAL TRIAL: NCT06430645
Title: Effects of Esketamine on Recovery of Consciousness After Propofol Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: esketamine_2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Post-anesthesia Recovery
MeSH Terms: interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose of esketamine (Experimental): Drug：esketamine (0.3mg/kg)
  Interventions: Drug: Esketamine
- high dose of esketamine (Experimental): Drug：esketamine(0.6mg/kg)
  Interventions: Drug: Esketamine
- control group (Experimental): Drug：0.9% saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esketamine — Sufentanil(0.1ug/kg) and flurbiprofen axetil(50mg) are administered before induction. Propofol (10 mg/ml) is infused via target-controlled infusions (TCIs). Esketamine hydrochloride (0.3mg/kg total body weight) single intravenous injection after stable plasma concentration of propofol deep sedation.
  Arms: low dose of esketamine
Drug: Esketamine — Sufentanil(0.1ug/kg) and flurbiprofen axetil(50mg) are administered before induction. Propofol (10 mg/ml) is infused via target-controlled infusions (TCIs). Esketamine hydrochloride (0.6mg/kg total body weight) single intravenous injection after stable plasma concentration of propofol deep sedation.
  Arms: high dose of esketamine
Drug: Saline — Sufentanil(0.1ug/kg) and flurbiprofen axetil(50mg) are administered before induction. Propofol (10 mg/ml) is infused via target-controlled infusions (TCIs). The same volume of 0.9% saline instead of esketamine will be given to the control group after stable plasma concentration of propofol deep sedation.
  Arms: control group

SUMMARY:
Esketamine is an antagonist of N-methyl-d-aspartate (NMDA) receptor different from other gamma-aminobutyric acid (GABA) receptor agonists. Recent studies showed that subanesthetic doses of ketamine not only deepen anesthesia but also accelerate recovery from isoflurane anesthesia in mice. It is necessary to verify if it applies to human. Besides inducing behavioral unresponsiveness, an optimal and important goal of general anesthesia is to prevent connected consciousness. The results of many studies support the conclusion that anesthesia-related unconsciousness is a consistent functional disconnection of lateral frontoparietal networks.The goal of this clinical trial is to learn if subanaesthetic doses of esketamine works to accelerate the recovery of consciousness from propofol anesthesia. It will also learn about the change of brain network when administrated the esketamine during propofol anesthesia. The main questions it aims to answer are:

1. Does subanaesthetic doses of esketamine can accelerate recovery from propofol anaesthesia?
2. What will happen to brain network connection after different doses of esketamine during propofol anesthesia?

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years to 50 years
* Patients scheduled for elective operative hysteroscopy
* Willing to sign informed consent

Exclusion Criteria:

* Contraindications of propofol and esketamine
* Contraindications for EEG;
* ASA≥III;
* BMI≥30 kg/m2 or BMI<18 kg/m2;
* The MMSE scale score is lower than the normal value;
* Alcohol or drug abuse;
* Untreated or under-treated hypertension, hyperthyroidism, risk of increased intracranial pressure, audio-visual impairment, history of psychiatric disorders or neurological diseases, malignant tumors or other major diseases;
* Use of other neurological drugs or drugs known to interact with propofol and esketamine in the past 2 weeks;
* Pregnant and lactating women;
* The operation duration is shorter than 15 minutes or longer than 60 minutes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery time | 2 hours
  Recovery time will be defined as the time from terminating propofol administration to opening eyes to verbal stimuli (participants addressed by name) or, if necessary, mild tactile stimuli (a tap in the shoulder) every 30 seconds.

SECONDARY OUTCOMES:
Explicit memory scores and implicit memory scores | 2 hours
  The task includes process-dissociation procedure with the word-stem completion. The value ranges from -1 to 1. If the value is less than or equal to 0, it means no memory. If the value is more than 0, it means memory is detected.
Subjective experience report | 2 hours
  The judges of structured interviews includes three main categories: reports of no recall of any experiences, white reports and reports with specific content.
Grooved Pegboard Test points | 2 hours
  Time to complete the Grooved Pegboard Test with dominant and non-dominant hand.
Patients state index | 2 hours
  Processed EEG will be recorded using Sedline (Masimo, Irvine, CA, USA). Patients state index (PSI) uses a proprietary algorithm that incorporates a combination of quantitative EEG parameters and ranges from 0 to 100, with 100 being associated with wakefulness and 0 with an isoelectric EEG.
Spectral edge frequency | 2 hours
  Spectral edge frequency (SEF) is calculated from the power in frequency ranges. The area under the curve of the power spectrum is calculated and the SEF95 is derived by calculating the frequency at which power is separated into 95 and 5%. SEF90 is calculated in a similar way.
Burst suppression ratio | 2 hours
  Burst-suppression ratio would be 1.0 for an isoelectric EEG signal and 0 for an EEG signal without any isoelectric periods and represents the percentage of the previous 63 seconds epoch of EEG recognized as those periods longer than 0.5 second, during which the EEG voltage does not exceed approximately +5 to - 5 μV, indicating a severe reduction in the brain's neuronal activity and metabolic rate.
Original EEG | 2 hours
  Four simultaneous channels of frontal EEG waveforms reflect electrical activity of the frontal and pre-frontal cortices of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China